CLINICAL TRIAL: NCT05741099
Title: The Application and Research of Mesenchymal Stem Cells in Alleviating the Severe Development of Novel Coronavirus Infection to Clarify Its Safety and Effectiveness.
Brief Title: Application and Research of Mesenchymal Stem Cells in Alleviating Severe Development of COVID-19 Infection
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Medical University (Other)
Responsible Party: Principal Investigator, Quanhai Li, Director of the Cell Therapy Laboratory, Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-MSCs-COVID-19
Record Dates: First submitted 2023-02-10; First posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: COVID-19
Keywords: MSC; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MSCs group (Experimental): Patient in Mscs group will receive MSCs implantation by intravenous injection Within 10-15 days of infection
  Interventions: Biological: Umbilical cord mesenchymal stem cells implantation
- comparator (Placebo Comparator): Patients in comparator group will receive placebo treatment Within 10-15 days of infection
  Interventions: Other: Comparator

INTERVENTIONS:
Biological: Umbilical cord mesenchymal stem cells implantation — Patient in Mscs group will receive MSCs implantation by intravenous injection.
  Arms: MSCs group
Other: Comparator — Patients in comparator group will receive placebo treatment
  Arms: comparator

SUMMARY:
This study is to evaluate the safety and efficacy of umbilical cord mesenchymal stem cells Therapy for COVID-19.

DETAILED DESCRIPTION:
Since 2019, novel coronavirus Disease 2019 (COVID-19) has spread and prevailed all over the world. COVID-19 has a wide range of clinical manifestations of respiratory and non-respiratory symptoms, including mild or severe influenza-like syndrome, respiratory distress or respiratory failure, and may end in multiple organ failure. Mesenchymal stem cells (MSCS) are considered as ideal seed cells for the treatment of various diseases due to their unique immune regulation, self-renewal and multiple differentiation potentials. The safety of MSC transplantation in the treatment of COVID-19 patients has been proved by a number of clinical studies, and has shown good clinical efficacy in shortening the course of the disease, alleviating lung damage, and reducing the level of inflammatory factors. However, previous clinical studies mainly focused on the efficacy of MSC transplantation in critically ill patients of COVID-19, ignoring the important role of cell transplantation in delaying or preventing COVID-19 's progress and preventing reinfection.COVID-19 has spread throughout the country and even the world, and the increase in severe and critical cases has caused a great impact on national medical and health resources. Stem cell transplantation offers new treatment ideas for COVID-19 patients. Since the role of cell transplantation in delaying or preventing the progression of light and medium novel coronavirus infection and preventing reinfection has not been clearly reported, this study intends to use MSC transplantation to evaluate the role of stem cells in the occurrence and development of novel coronavirus infection, so as to provide an important reference for the prevention and treatment of COVID-19 by MSC.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85 years;The diagnosis of COVID-19 infection was clinically classified as Moderate cases, and the criteria were based on Diagnosis and Treatment Protocol for Novel Coronavirus Pneumonia(Trial Version 10)
* Having the relevant clinical manifestations of COVID-19 infection.
* Having one or more of the following etiological and serological examination results
* Tested positive for Novel Coronavirus nucleic acid
* Tested positive for Novel Coronavirus antigen
* Novel Coronavirus was isolated and cultured positive
* Novel Coronavirus specific immunoglobulin G reaches a titration of at least 4-fold increase during convalescence compared with the acute phase.
* Moderate cases diagnostic criteria：Persistent high fever > 3 days or (and) cough, Tachypnea etc，but respiratory rate≧30 breaths/ min ,oxygen saturation > 93% on finger pulse oximeter taken at rest. Radiology shows the characteristic manifestations of COVID-19 pneumonia
* There are one or more of the following risk factors for the development of severe / critical severity:
* Patients over 65 years old, especially those who have not been vaccinated against novel coronavirus
* Patients with cardiovascular and cerebrovascular diseases (including hypertension), chronic lung disease, diabetes, chronic liver and kidney disease, tumors and other underlying diseases, as well as maintenance dialysis
* Patients with immune deficiency (such as AIDS, long-term use of corticosteroids or other immunosuppressive drugs resulting in immune dysfunction)
* Patients with Obesity (body mass index ≥30)
* late trimester of pregnancy and perinatal women
* Heavy smoker.

Exclusion Criteria:

* Patients with prior or present tumor history,or precancerous lesions confirmed by pathological examination.
* Patients with active acute myocardial infarction or acute cerebral infarction.
* Pregnant or lactating patients.
* Patients with poorly controlled mental illness.
* Patients addicted to alcohol or drugs.
* Patients Unable or unwilling to sign informed consent or poor compliance.
* Patients with active tuberculosis or influenza virus, adenovirus and other acute respiratory virus infection.
* Patients deemed unsuitable for stem cell therapy by clinicians.
* Patients enrolled in other clinical trials within 3 months.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-01-28 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Effectiveness evaluation | Within 1 year of receiving mesenchymal stem cell transplants
  The incidence and clinical status of progression to critical type after the third stem cell transplantation were evaluated

SECONDARY OUTCOMES:
Hospitalization time | Time period from patient admission to discharge
  The patient's hospital stay in days should be recorded.
oxygenation index（OI） | At the time of our patient's hospitalization and 7 days after receiving the third MSC transplant.
  The oxygenation index of the patient was quantitatively measured in mmHg.
Oxygen saturation（SaO2） | At the time of our patient's hospitalization and 7 days after receiving the third MSC transplant.
  The blood oxygen saturation of patients was monitored by oximeter.
Chest CT | At admission, before to the stem cell transplant, and at 1 month, 6 months, and 12 months following the third MSC transplant.
  A computed tomography (CT) scan of the patient's chest was performed to evaluate the level of inflammation, the scope of the involvement, and the degree of fibrosis in the heart and lungs.
Pulmonary function evaluation | At admission, before to the stem cell transplant, and at 1 month, 6 months, and 12 months following the third MSC transplant.
  Lung ventilation experiments were used to measure the lung volume (in ml) and airway patency (in ml) of patients in order to assess their lung function.
Blood biochemical examination | At admission, before to the stem cell transplant, and at 1 month, 6 months, and 12 months following the third MSC transplant.
  The progression of the lesion was determined by blood chemistry tests on a patient's blood sample, which mostly included liver function: Alanine aminotransferase (U/L)，Glutamic oxaloacetic transaminase (U/L), renal function:blood urea nitrogen (mmol/L) and serum creatinine (umol/L), cardiac function: creatine kinase isoenzymes(U/L) and Troponin(ng/ml), and inflammatory factors: C- reactive protein (mg/dl) and Interleukin- 6(Pg/ml) .
Echocardiographic examination of heart function | At admission, before to the stem cell transplant, and at 1 month, 6 months, and 12 months following the third MSC transplant.
  Echocardiography was used to evaluate the patient's myocardial contractility, primarily focusing on left ventricular ejection fraction (LVEF).
Safety assessment | Within 1 year of receiving mesenchymal stem cell transplants
  infusion and allergic reactions, life-threatening adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Xifeng Jiang, Doctor, Study Chair — The First Hospital of Hebei Medical University; Gang Liu, Master, Study Director — The First Hospital of Hebei Medical University; Wuzhuang Sun, Master, Study Director — The First Hospital of Hebei Medical University; Baoyong Yan, Master, Principal Investigator — The First Hospital of Hebei Medical University; Mingqi Zheng, Master, Principal Investigator — The First Hospital of Hebei Medical University; Ding Yu, Master, Principal Investigator — The First Hospital of Hebei Medical University; Le Wang, Master, Principal Investigator — The First Hospital of Hebei Medical University; Yajie Wang, Master, Principal Investigator — The First Hospital of Hebei Medical University; Quanhai Li, Master, Principal Investigator — The First Hospital of Hebei Medical University; Xianyun Wang, Doctor, Principal Investigator — The First Hospital of Hebei Medical University; Jiawei Yang, Postgraduate, Principal Investigator — The First Hospital of Hebei Medical University; Tianshuo Li, Postgraduate, Principal Investigator — The First Hospital of Hebei Medical University
Locations (1):
- The First Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Munster VJ, Koopmans M, van Doremalen N, van Riel D, de Wit E. A Novel Coronavirus Emerging in China - Key Questions for Impact Assessment. N Engl J Med. 2020 Feb 20;382(8):692-694. doi: 10.1056/NEJMp2000929. Epub 2020 Jan 24. No abstract available. PMID 31978293
- [Result] Galipeau J, Sensebe L. Mesenchymal Stromal Cells: Clinical Challenges and Therapeutic Opportunities. Cell Stem Cell. 2018 Jun 1;22(6):824-833. doi: 10.1016/j.stem.2018.05.004. PMID 29859173
- [Result] Hashemian SR, Aliannejad R, Zarrabi M, Soleimani M, Vosough M, Hosseini SE, Hossieni H, Keshel SH, Naderpour Z, Hajizadeh-Saffar E, Shajareh E, Jamaati H, Soufi-Zomorrod M, Khavandgar N, Alemi H, Karimi A, Pak N, Rouzbahani NH, Nouri M, Sorouri M, Kashani L, Madani H, Aghdami N, Vasei M, Baharvand H. Mesenchymal stem cells derived from perinatal tissues for treatment of critically ill COVID-19-induced ARDS patients: a case series. Stem Cell Res Ther. 2021 Jan 29;12(1):91. doi: 10.1186/s13287-021-02165-4. PMID 33514427
- [Result] Zanirati G, Provenzi L, Libermann LL, Bizotto SC, Ghilardi IM, Marinowic DR, Shetty AK, Da Costa JC. Stem cell-based therapy for COVID-19 and ARDS: a systematic review. NPJ Regen Med. 2021 Nov 8;6(1):73. doi: 10.1038/s41536-021-00181-9. PMID 34750382
- [Result] Wang C, Horby PW, Hayden FG, Gao GF. A novel coronavirus outbreak of global health concern. Lancet. 2020 Feb 15;395(10223):470-473. doi: 10.1016/S0140-6736(20)30185-9. Epub 2020 Jan 24. No abstract available. PMID 31986257
- [Result] Xu Z, Shi L, Wang Y, Zhang J, Huang L, Zhang C, Liu S, Zhao P, Liu H, Zhu L, Tai Y, Bai C, Gao T, Song J, Xia P, Dong J, Zhao J, Wang FS. Pathological findings of COVID-19 associated with acute respiratory distress syndrome. Lancet Respir Med. 2020 Apr;8(4):420-422. doi: 10.1016/S2213-2600(20)30076-X. Epub 2020 Feb 18. No abstract available. PMID 32085846
- [Result] Wang Y, Chen X, Cao W, Shi Y. Plasticity of mesenchymal stem cells in immunomodulation: pathological and therapeutic implications. Nat Immunol. 2014 Nov;15(11):1009-16. doi: 10.1038/ni.3002. PMID 25329189
- [Result] Leng Z, Zhu R, Hou W, Feng Y, Yang Y, Han Q, Shan G, Meng F, Du D, Wang S, Fan J, Wang W, Deng L, Shi H, Li H, Hu Z, Zhang F, Gao J, Liu H, Li X, Zhao Y, Yin K, He X, Gao Z, Wang Y, Yang B, Jin R, Stambler I, Lim LW, Su H, Moskalev A, Cano A, Chakrabarti S, Min KJ, Ellison-Hughes G, Caruso C, Jin K, Zhao RC. Transplantation of ACE2- Mesenchymal Stem Cells Improves the Outcome of Patients with COVID-19 Pneumonia. Aging Dis. 2020 Mar 9;11(2):216-228. doi: 10.14336/AD.2020.0228. eCollection 2020 Apr. PMID 32257537
- [Result] Shu L, Niu C, Li R, Huang T, Wang Y, Huang M, Ji N, Zheng Y, Chen X, Shi L, Wu M, Deng K, Wei J, Wang X, Cao Y, Yan J, Feng G. Treatment of severe COVID-19 with human umbilical cord mesenchymal stem cells. Stem Cell Res Ther. 2020 Aug 18;11(1):361. doi: 10.1186/s13287-020-01875-5. PMID 32811531